CLINICAL TRIAL: NCT04782414
Title: Observational Study of Patients Treated With Hot AXIOS® Prosthesis in Real Life Conditions -
Brief Title: Hot AXIOS® Prosthesis in Real Life Conditions -
Acronym: REALAXIOS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-PP-20
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pancreatitis,Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hot AXIOS® prosthesis — endoscopic trans digestive drainage using of the Hot AXIOS prosthesis in the treatment of pancreatic collections (incompletely fluid or necrotic)

SUMMARY:
Regulatory Context The CNEDiMTS makes the renewal of registration conditional on the transmission of the results of a well-conducted prospective study, carried out with Hot AXIOS, the objective of which is to evaluate the interest of this device in real conditions of use with regard to effectiveness and complications after a minimum follow-up of 3 months.

Operators are trained in the use of the equipment (practice on ex-vivo model and/or prior stent placement) and undertake to comply with the rules and formalities of use.

Primary efficacy objective :

To evaluate the efficacy of endoscopic trans digestive drainage after use of the Hot AXIOS prosthesis in the treatment of pancreatic collections (incompletely fluid or necrotic) at 3 months.

Secondary Objectives :

Assessment of the following elements :

1. Morbidity (complication rates) and mortality per- and post-procedure
2. Recurrence rate of pancreatic collection
3. Evolution of the quality of life questionnaire (SQ5D5L)
4. Technical success rate of prosthesis placement and removal success rate of the prosthesis
5. Search for factors predictive of clinical success of endoscopic pancreatic drainage with the Hot Axios prosthesis.

Study design Non-interventional/observational (RIPH 3 type), multi-center, prospective study with consecutive inclusions evaluating the Hot AXIOS® prosthetic device.

Non-inclusion registry A minimum amount of information will be collected anonymously, including sex, age, indication of drainage and reason for non-inclusion (e.g. refusal of the patient, of the investigator for impossibility of following the patient in the centre or other reasons to be specified). Generic information will be affixed in each centre participating in the study indicating: "In application of the provisions of the Data Protection Act, general information on the possibility that personal data may be used for research purposes must be provided in any establishment or centre where prevention, diagnosis and care activities are carried out". This must be exhaustive and rigorously maintained.

Equipment used in endoscopy Hot AXIOS™ - self-expanding metal prosthesis with a lumen diameter of 6 to 20 mm and collar length of 8 and 10 mm or any future similar device marketed under the same name at the time of the study.

Technique Insertion of the material under echo-endoscopic control -- possible but not systematic dilatation -- guide wire with hydrophilic tip - Puncture and release under echo-endoscopic control according to the centre's usual practice.

Registration The data will be collected anonymously in an electronic computer database using eCRFs.

Statistical analysis The evaluation of the clinical success of endoscopic pancreatic necrosectomy with metallic prosthesis will first consist in describing its efficacy according to the criteria described above.

Analysis plan :

The statistical analysis will first include a description of the study population with the number of patients falling under the indication and treated with the Hot AXIOS system at the recruiting centers (source population), the number of eligible patients who consented to participate in the study, the number of patients included (study population), the number of subjects who made each visit and were analyzed, premature exits (deaths, lost to follow-up) will be reported and described in the form of a flow chart.

ELIGIBILITY:
Inclusion Criteria:

* Should benefit from the installation of a Hot Axios system as part of PBDA support, regardless of the indication.
* Age ≥ 18 years old,
* Having signed his or her no objection or the trusted person if the patient is unable to do so prior to the procedure
* Affiliated to a social security scheme

Exclusion Criteria:

• Patients who have indicated that they do not wish to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having benefited from the treatment of pancreatic collections
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
patients with clinical success | 3 months
  reduction in the size of the pancreatic fluid collection ≤ 3 cm, evaluated by imaging

SECONDARY OUTCOMES:
Collect all complications, | 3 months
  Complications will be assessed according to Cotton's endoscopic classification26 (mild, moderate, severe, or fatal) [Cotton PB, Eisen GM, Aabakken L, et al. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc.2010; 71: 446-54].
recurrence of pancreatic collection | 3 months
  the presence of a collection of pancreatic origin on imaging of more than 3 cm at the 3-month check-up
evolution of the quality of life questionnaire | 3 months
  Analyze the evolution of the quality of life questionnaire EQ5D5L, with as reference the one completed before the procedure
Evaluate the technical success rate | 3 months
  success of the prosthesis in place at the end of the endoscopic procedure - determined by the correct trans parietal (gastric or duodenal) deployment (collar on either side of the digestive walls) and the technical success rate of the prosthesis removal (endoscopic extraction) and the date of the procedure.
Look for factors predictive of clinical success | 3 months
  the predictive factors will be an aggregate of the folowing clinicals signs
  1. sex, age, body mass index, severity score (APACHE II), aetiology of pancreatitis, size of collection, proportion of solid debris in the collection, associated pancreatic ductal rupture, glandular extension and peritoneal extension of the necrosis , location of the gastrostomy , time between admission and completion of the procedure
  2. According to the clinical signs that motivated the intervention such as :
  i. Pain and/or, ii. Necrosis infection (positive culture of necrosis, presence of gas bubbles in the collection on imaging, persistent sepsis or deterioration of the patient's condition malgré́ an optimal resuscitation support without documented infection) and/or, iii. High occlusion (vomiting, food intolerance and gastric stasis on imaging) and/or, iv. Symptoms such as jaundice and/or, v. Organ failures such as kidney, heart, lung.

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Avignon Hospital, Avignon
  - brest Hospital, Brest
  - Clermont-ferrand hospital, Clermont-Ferrand
  - Polyclinique Saint Côme, Compiègne
  - Lille Hospital, Lille
  - Limoges hospital, Limoges
  - Clinique Jean Mermoz, Lyon
  - APHM, Marseille
  - European Hospital, Marseille
  - St Joseph Hospital, Marseille
  - Nancy Hospital, Nancy
  - Nice Hospital, Nice
  - APHP saint antoine, Paris
  - Hôpital privé des peupliers, Paris
  - Poitiers Hospital, Poitiers
  - Saint Etienne Hospital, Saint-Etienne
  - Centre Hospitalier Jacques Lacarin, Vichy

IPD SHARING:
Plan to Share IPD: No